CLINICAL TRIAL: NCT04088760
Title: Safety and Efficacy of TCRαβ+/CD19+ Depleted Allogeneic Hematopoietic Stem Cell Transplantation for Malignant and Non-malignant Disorders in Children and Adolescent/Young Adult Patients
Brief Title: TCRαβ+/CD19+ Depleted Allogeneic Hematopoietic Stem Cell Transplantation for Malignant and Non-malignant Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Post-transplant cyclophosphamide and abatacept can be used as standard-of-care approaches to GVHD prevention in the HLA mismatched donor-recipient setting and are simpler to use since study enrollment is not required.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-8568
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Allogeneic Hematopoietic Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TCRαβ+/CD19+ depleted HSCT (Experimental)
  Interventions: Drug: TCRαβ+/CD19+ depleted allogeneic hematopoietic stem cell transplant (HSCT)

INTERVENTIONS:
Drug: TCRαβ+/CD19+ depleted allogeneic hematopoietic stem cell transplant (HSCT) — The majority of TCRαβ+ T cells and CD19+ B cells will be removed from the allogeneic graft utilizing the CliniMACS® immunomagnetic selection device (Miltenyi Biotec). The depletion process involves two phases; cell labeling (phase 1) and the automated immunomagnetic depletion process (phase 2). The CD34+ dose may be adjusted by the need to not exceed the TCRαβ+CD3+ dose threshold.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of TCRαβ+/CD19+ depleted allogeneic hematopoietic stem cell transplant (HSCT) for malignant and non-malignant disorders in children and adolescent/young adult patients using the CliniMACS® immunomagnetic selection device (Miltenyi Biotec).

DETAILED DESCRIPTION:
Acute graft versus host disease (GVHD) remains a significant cause of morbidity and mortality and is the biggest barrier to successful allogeneic hematopoietic cell transplantation (HSCT) outcomes. Improved methods of acute GVHD prevention are needed. TCRαβ+/CD19+ depletion of allogeneic hematopoietic stem cell products offers an opportunity to limit the risk of acute GVHD by removing TCRαβ+ T cells and CD19+ B cells which participate in acute GVHD initiation and perpetuation. The purpose of this study is to investigate the safety and efficacy of TCRαβ+/CD19+ depleted allogeneic hematopoietic stem cell transplant (HSCT) for malignant and non-malignant disorders in children and adolescent/young adult patients using the CliniMACS® immunomagnetic selection device (Miltenyi Biotec).

ELIGIBILITY:
Inclusion Criteria:

* Any patient being treated at Cincinnati Children's Hospital requiring an allogeneic HSCT who lacks an HLA-genotypically matched related donor. Genotypically matched related donors are allowed when there is a clinical desire to avoid the use of GVHD prophylaxis medications.

Exclusion Criteria:

* Prior allogeneic transplant with active acute or chronic GVHD, or life-threatening infection. Patients with a prior history of allogenic transplant without active GVHD or life-threatening infection can be considered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TCRαβ+/CD19+ Depleted HSCT
Started | 15
Completed | 14
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | TCRαβ+/CD19+ Depleted HSCT
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Caucasian | 7
  Hispanic | 4
  African American | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Infusion-related Reactions
Description: Number of patients who experienced infusion reactions including rash, fever, difficulty breathing, and blood pressure abnormalities at the time of infusion of stem cells.
Time Frame: 100 days
Measure: Number; unit: number of infusion reactions
Units Other Than Participants: infusions
Arm/Group | TCRαβ+/CD19+ Depleted HSCT
Number analyzed (Participants) | 14
Number analyzed (infusions) | 16
number of infusion reactions | 1

2. Secondary Outcome: Engraftment and Sustained Donor Chimerism
Description: Initial neutrophil engraftment prior to day +28 was determined by monitoring for neutrophil count recovery post-transplant and performing blood tests to confirm presence of donor cells. Sustained donor chimerism at 1 year post transplant was determined again by performing blood tests to confirm presence of donor cells.
Time Frame: 28 days and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TCRαβ+/CD19+ Depleted HSCT
Number analyzed (Participants) | 14
Participants
  Neutrophil Engraftment | 13
  Sustained donor engraftment at 1 year | 5

3. Secondary Outcome: Number of Participants With Acute GVHD
Description: Patients were monitored for symptoms of acute graft versus host disease including rash, diarrhea, and increased bilirubin using the Modified Glucksberg Criteria.
Time Frame: 100 days
Population: 14 patients received 15 transplants.
Measure: Count of Participants; unit: Participants
Arm/Group | TCRαβ+/CD19+ Depleted HSCT
Number analyzed (Participants) | 14
Participants | 5

4. Secondary Outcome: Number of Participants With Chronic GVHD
Description: Patients were monitored for symptoms of chronic graft versus host disease using the NIH Consensus Criteria.
Time Frame: 1 year
Population: Five patients were evaluable for chronic graft versus host disease at 1 year time point.
Measure: Count of Participants; unit: Participants
Arm/Group | TCRαβ+/CD19+ Depleted HSCT
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: GVHD-free Survival
Description: GVHD-free survival was determined based on the presence or not of acute or chronic GVHD at 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TCRαβ+/CD19+ Depleted HSCT
Number analyzed (Participants) | 11
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the first week of the study. Serious Adverse Events and All-Cause Mortality were collected up to 1 year.
Description: Only events that were determined to be attributable to study intervention noted after the first week were recorded and reported.
Arm/Group | TCRαβ+/CD19+ Depleted HSCT
All-Cause Mortality (participants affected / at risk) | 6/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCRαβ+/CD19+ Depleted HSCT (N=15)
Sepsis (Infections and infestations) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCRαβ+/CD19+ Depleted HSCT (N=15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Worsening pain (General disorders) | 3 (3)
Hypokalemia (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Bacteremia (strep mitis) (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT04088760/Prot_SAP_000.pdf